CLINICAL TRIAL: NCT02884609
Title: Tolerance and Efficiency of Paracetamol bu Subcutaneous Releasing in Patients Hospitalized Into Palliative Care
Brief Title: Tolerance and Efficiency of Paracetamol Subcutaneous Injection
Acronym: TEPASC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-02Obs-CHRMT
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2016-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the tolerance and the efficiency of subcutaneous administration of Paracetamol for patients in palliative care.

DETAILED DESCRIPTION:
Subcutaneous administration is the most commonly used way for palliative care and geriatric service. A lot of drugs are recommended with subcutaneous administration, but their use is performed out of the Marketing Authorization, and fewer data exist about this practice in literature. Paracetamol is a grade 1 analgesic not currently recommended for subcutaneous injection, because of the lack of validated references. However this kind of administration is usually performed for Paracetamol in the French palliative care services related with its advantages for patients, as analgesic or antipyretic. The assumption of the study is that the use of paracetamol subcutaneously is possible with a good tolerance for hospitalized patients in palliative care service.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years old
* indication of paracetamol by subcutaneous injection, as an analgesic or an antipyretic

Exclusion Criteria:

* opposition to gather data patient
* subcutaneous administration of paracetamol during the last week before the inclusion of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in palliative care service with an indication of Paracetamol by subcutaneous injection
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2014-08; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of the severe or not adverse effects on the injection site | 8 days

SECONDARY OUTCOMES:
as antipyretic, a feedback of tympanic temperature below 38°C during the two hours after injection | 8 days
as analgesic, the decrease of pain (decrease of 30 in the numerical scale score, or a Algo+ scale score lower than 2/5) | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Benoît LEHEUP, MD, Principal Investigator — CHR Metz-Thionville
Locations (2):
- France (2):
  - CHR Metz-Thionville, Metz
  - GH Diaconesses Croix Saint Simon, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leheup BF, Ducousso S, Picard S, Alluin R, Goetz C. Subcutaneous administration of paracetamol-Good local tolerability in palliative care patients: An observational study. Palliat Med. 2018 Jul;32(7):1216-1221. doi: 10.1177/0269216318772472. Epub 2018 May 8. PMID 29737243